CLINICAL TRIAL: NCT02147314
Title: Evaluation of the YOFiLife Blood Glucose Monitoring System With YOFiMeter Glucometer
Brief Title: Evaluation of the YOFiMeter Glucometer
Status: Completed | Type: Observational
Sponsor: YofiMeter, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: YOFiMeter 2013-1
Record Dates: First submitted 2014-05-21; First posted 2014-05-26 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes
Keywords: diabetes; glucometer; Yofimeter; diabetes monitoring
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This evaluation will evaluate a new system from YOFiMeter, known as YOFiLife Blood Glucose Monitoring System with YOFiMeter glucometer. YOFiLife includes a web- based data system known as the Web Portal and smart phone apps for the iPhone and Android. The new YOFiMeter is similar to other glucometers with the exception of built in test cassettes, lancet cassettes with enhanced communications and data reviewing options.

This evaluation will also collect data from a YSI 2300 Stat Plus Glucose Analyzer reference glucometer. The YSI 2300 Stat Plus Glucose Analyzer will be used as the "gold" standard with all results compared to the YSI results.

DETAILED DESCRIPTION:
This is a single evaluation to assess both the Yofimeter system accuracy in the hands of the intended users, as well as other aspects to support lay use, such as labeling assessment and usability. The company is presenting diabetics who monitor their blood glucose with new technological innovations aimed at improving their daily lives (e.g., a unique blood glucose monitor, Web Portal applications and "smart phone" applications).

Each subject selected for the comparison evaluation will perform their own fingerstick and test on their subject device following device instructions. A trained technician will perform a fingerstick on the subject immediately after and perform the test on the same device. Separate results will be recorded by subject and technician. A trained technician will take another blood sample, within as short of a time as practicable, for a glucose assay on the YSI 2300 Stat Plus Glucose Analyzer.

ELIGIBILITY:
Inclusion Criteria:

1. Is the subject currently self-testing for blood glucose levels?
2. Is the subject able to provide legal, written informed consent?
3. Is the subject willing to have fingersticks for blood glucose determination?
4. Does the subject show an ability and willingness to follow directions of the Investigator and staff?
5. Is the subject 18 years of age or older?
6. Does the subject have a hematocrit value in the range of 20-60?

Exclusion Criteria:

1. Does the subject demonstrate a lack of compliance as determined by the Principal or Lead Site Investigator and/or staff?
2. Is the subject currently participating in another clinical study of an investigational device or drug?
3. Is the subject unwilling or unable to provide concurrent blood glucose level determinations with the YOFiMeter whenever blood glucose levels are determined at the Investigator's site?
4. Is the subject, or a family member, employed by a company that develops or markets blood glucose level determining devices?
5. Does the subject have any other condition or finding, which in the opinion of the investigator would make the subject unsuitable for enrollment, or could interfere with the subject participating in and completing the protocol?
6. Is the subject unwilling or unable to provide Informed Consent (IC)?

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals over 18 years of age with diabetes who currently use blood glucose monitors.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Accuracy of the Yofimeter as compared to the YSI 2300 Stat Plus Glucose Analyzer | Within the hour
  The patient- and provider- measures of blood glucose will be compared to the YSI Analyzer measures using the standard statistical methods for method-validation analysis: Bland-Altman agreement and Passing-Bablok regression.

SECONDARY OUTCOMES:
Evaluate the usability of instructional materials. | Within 2 hours
  Evaluate the usability of the instructional materials in assisting a new user to set up and use the YOFiLife Blood Glucose Meter and the data monitoring systems, on the Web Portal, and mobile iPhone and Android apps.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bailey, MD, Principal Investigator — AMCR Institute
Locations (3):
- United States (3):
  - Profil Institute for Clinical Research, Chula Vista, California
  - AMCR Institute, Escondido, California
  - Tri City Endocrinology, Oceanside, California